CLINICAL TRIAL: NCT05446441
Title: Endoscopic Thyroidectomy Using Gasless Unilateral Transaxillary Approach Versus Conventional Open Thyroidectomy for Papillary Thyroid Cancer: a Prospective, Multicenter, Randomized Controlled Clinical Trial
Brief Title: Endoscopic Thyroidectomy Versus Open Thyroidectomy for Papillary Thyroid Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Minghua Ge, PH.D, Zhejiang Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022（050）
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; Endoscopic surgery; Open surgery; Radical thyroidectomy
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention; (Experimental): Endoscopic thyroidectomy was performed in a standardized fashion by multi-institutional Chinese experienced surgeons using the same gasless unilateral transaxillary approach.
  Interventions: Procedure: Endoscopic surgery;
- Control (Active Comparator): Conventional open surgery was performed in a standardized fashion by multi-institutional Chinese experienced surgeons.
  Interventions: Procedure: Endoscopic surgery;

INTERVENTIONS:
Procedure: Endoscopic surgery; — Endoscopic thyroidectomy group is the papillary thyroid carcinoma patient group who underwent endoscopic thyroid surgery using a gasless, trans-axillary approach.

SUMMARY:
Recently, endoscopic thyroidectomy using gasless unilateral transaxillary approach has been proven feasible and safe in several Chinese medical centers. This study is aimed to compare multi-institutional Chinese outcomes of endoscopic thyroidectomy using gasless unilateral transaxillary approach and conventional open surgery.

DETAILED DESCRIPTION:
Most patients with thyroid tumors are effectively treated surgically by practitioners experienced in the techniques of thyroidectomy. Many patients, especially women, undergoing thyroid surgery are concerned about the postoperative cosmetic appearance of the neck. Endoscopic thyroidectomy using gasless unilateral transaxillary approach which can hide the operative scar was associated with a higher degree of patient cosmetic satisfaction. Recently, endoscopic thyroidectomy using gasless unilateral transaxillary approach has been proven feasible and safe in several Chinese medical centers. In this study, we designed a prospective study comparing multi-institutional Chinese outcomes of endoscopic thyroidectomy using gasless unilateral transaxillary approach and conventional open surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* The pathological type is papillary thyroid carcinoma;
* Tumor diameter <2 cm；
* No extraglandular invasion, or minimal extrathyroidal extension invading only anterior thyroid capsule or sternothyoid muscle；
* cN0 or cN+ without fusion and fixation of metastatic lymph nodes；
* no obvious contraindication for thyroidectomy ;
* Good comply with the research visit plan and other program requirements;
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* patients with severe systemic diseases who can not tolerate general anesthesia or routine surgical posture;
* previous history of neck surgery, radiotherapy or thermal ablation;
* hyperthyroidism and substernal goiter;
* dedifferentiated thyroid carcinoma；
* accompanied with severe thyroiditis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Estimated)
Dates: Start 2022-06-28 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of retrieved central lymph nodes | 1 month after operation
  The number of central lymph nodes removed during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Minghua Ge, Doctor, Principal Investigator — Zhejiang Provincial People's Hospital

IPD SHARING:
Plan to Share IPD: No